CLINICAL TRIAL: NCT00518895
Title: A Multicenter, Randomized, Double-blind Study of Dacarbazine With or Without Genasense in Chemotherapy-naive Subjects With Advanced Melanoma and Low LDH (The AGENDA Trial)
Brief Title: Trial of Dacarbazine With or Without Genasense in Advanced Melanoma
Acronym: AGENDA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genta Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AGENDA; GM307
Record Dates: First submitted 2007-08-14; First posted 2007-08-21 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2009-04

CONDITIONS: Melanoma
Keywords: Melanoma; Advanced Melanoma; Malignant Melanoma; Metastatic Melanoma; Skin Cancer; Genasense; oblimersen; antisense; Bcl-2 antisense; G3139; dacarbazine
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — Dacarbazine; oblimersen; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Dacarbazine with Genasense
  Interventions: Drug: dacarbazine plus Genasense
- B (Active Comparator): Dacarbazine with placebo
  Interventions: Drug: dacarbazine plus placebo

INTERVENTIONS:
Drug: dacarbazine plus Genasense — Protocol therapy will be administered in 21-day cycles for up to 8 cycles. Subjects in the dacarbazine plus Genasense group will receive Genasense 7 mg/kg/day by continuous intravenous infusion beginning on Day 1 and continuing for 5 days (120 hours) plus dacarbazine 1000 mg/m2 as a 60-minute intravenous infusion immediately following the conclusion of the Genasense infusion. Subjects who are responding or have stable disease after 8 cycles of therapy may, at the Investigator's discretion, continue that same therapy for up to 8 additional cycles.
  Other Names: dacarbazine plus Genasense (oblimersen, G3139)
  Arms: A
Drug: dacarbazine plus placebo — Protocol therapy will be administered in 21-day cycles for up to 8 cycles. Subjects in the dacarbazine plus placebo group will receive placebo (that is, locally available commercial 0.9% Sodium Chloride Injection) by continuous intravenous infusion beginning on Day 1 and continuing for 5 days (120 hours) plus dacarbazine 1000 mg/m2 as a 60-minute intravenous infusion immediately following the conclusion of the placebo infusion. Subjects who are responding or have stable disease after 8 cycles of therapy may, at the Investigator's discretion, continue that same therapy for up to 8 additional cycles.
  Other Names: dacarbazine plus placebo (0.9% Sodium Chloride Injection)
  Arms: B

SUMMARY:
This study is being performed to prospectively determine whether dacarbazine plus Genasense is significantly better than dacarbazine plus placebo in chemotherapy-naive patients with advanced melanoma and low baseline LDH (LDH less than or equal to 0.8 times the upper limit of normal). LDH is a biomarker strongly associated with improved outcomes in a recent trial of dacarbazine plus Genasense.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of melanoma
* Progressive disease that is not surgically resectable, or metastatic Stage IV
* Low-normal LDH, defined as ≤ 0.8 times the upper limit of normal
* No prior chemotherapy
* Measurable disease
* ECOG performance status ≤ 1
* At least 4 weeks and recovery from effects of major prior surgery or other therapy, including immunotherapy, radiation therapy, or cytokine, biologic or vaccine therapy
* Prior immunotherapy allowed
* Adequate organ function

Exclusion Criteria:

* Prior cytotoxic chemotherapy, including regional perfusion, or prior Genasense treatment
* Primary ocular or mucosal melanoma
* Bone-only metastatic disease
* History or presence of brain metastasis or leptomeningeal disease
* Significant medical disease other than cancer
* Organ allograft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2007-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Progression-free survival and overall survival | Every 42 days from date of randomization during protocol therapy

SECONDARY OUTCOMES:
Response rate, durable response rate, duration of response, safety | Response and progression every 42 days from date of randomization during protocol therapy

CONTACTS AND LOCATIONS:
Locations (77):
- United States (14):
  - University of South Alabama Hospital, Mitchell Cancer Institute, Mobile, Alabama
  - San Diego Pacific Oncology and Hematology Associates Inc., Encinitas, California
  - Redwood Regional Medical Group, Inc., Santa Rosa, California
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Hematology Oncology Centers of the Northern Rockies, Billings, Montana
  - Morristown Memorial - Atlantic Healthcare System, Morristown, New Jersey
  - Cancer Care Associates, Oklahoma City, Oklahoma
  - Cancer Care Associates, Site 1, Tulsa, Oklahoma
  - St. Luke's Cancer Center, Bethlehem, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - The West Clinic, Memphis, Tennessee
  - Texas Oncology - Sammons Cancer Center, Dallas, Texas
  - MD Anderson Cancer Center at University of Texas, Houston, Texas
- Australia (3):
  - Sydney Cancer Center, Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Westmead Hospital, Westmead, New South Wales
- Austria (3):
  - Universitatsklinik fur Dermatologie und Venerologie, Medizinische Universitat Innsbruck, Innsbruck
  - Landesklinikum St. Polten, Sankt Pölten
  - Medical University of Vienna, Vienna General Hospital, Vienna
- Canada (2):
  - London Regional Cancer Program, London, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
- Charles University, Dermatology Department, Prague, Czechia
- France (16):
  - CHU Saint Jacques, Besançon
  - Hopital Saint-Andre, Bordeaux
  - CHU Ambroise Pare, Boulogne-Billancourt
  - CHU Hotel Dieu, Clermont-Ferrand
  - CHU de Dijon, Hopital du Bocage Sud, Dijon
  - CHU de Grenoble, Hopital Albert Michallon, Grenoble
  - Centre Hospitalier du Mans, Le Mans
  - CHRU de Lille, Hopital Claude Huriez, Lille
  - Hopital de l'Hotel Dieu, Lyon
  - Hopital Sainte Marguerite, Marseille
  - Hopital Saint Eloi, Montpellier
  - CHU Hotel Dieu, Nantes
  - Hopital Saint-Louis, Paris
  - Hopital Robert Debre, Reims
  - CHU CH Nicolle, Rouen
  - Institut Gustave Roussy, Villejuif
- Germany (20):
  - Charite Universitatsmedizin Berlin, Berlin
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Vivantes Klinikum Neukoln, Klinik fur Dermatologie und Venerologie, Berlin
  - Klinik fur Dermatologie und Allergologie der Ruhr-Universitat Bochum, Bochum
  - Klinik und Poliklinik fur Dermatologie und Venerologie, Cologne
  - Helios Klinikum Erfurt, Erfurt
  - Klinik fur Dermatologie, Allergologie und Venerologie, Universitatsklinikum Essen, Essen
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Hautklinik Linden, Hanover
  - Klinikum der Friedrich-Schiller-Universitat Jena, Jena
  - Universitatklinikum A. o. R., Leipzig
  - Hospital of the University of Schleswig-Holstein, Lübeck
  - Universitats-Hautklinik Mainz, Mainz
  - Universitatsklinikum Mannheim, Mannheim
  - Universitatsklinikum Giessen und Marburg GmbH, Klinik fur Dermatologie und Allergologie, Marburg
  - Klinik und Poliklinik fur Hautkrankheiten, Münster
  - Helios Vogtland-Klinikum Plauen, Plauen
  - Klinikum Quedlinburg, Quedlinburg
  - Dermatologische Klinik und Poliklinik, Regensburg
  - Hautklinik Universitat Tubingen, Tübingen
- Italy (6):
  - Ospedale San Salvatore, Coppitto-L'Aquila
  - Istituto Nazionale dei Tumori, Milan
  - Istituto Nazionale dei Tumori "G. Pascale", Napoli
  - IFO Instituto Regina-Elena - IRCCS, Rome
  - Istituto Dermopatico dell'Immacolata, Rome
  - Azienda Ospedaliera Universitaria di Siena, Siena
- Poland (2):
  - Szpital Akademii Medycznej w Gdansku, Gdansk
  - Wielkopolskie Centrum Onkologii, Poznan
- Spain (4):
  - Hospital Clinic I Provincial de Barcelona, Barcelona
  - Hospital Germans Trias I Pujol, Barcelona
  - Hospital Gregorio Maranon, Madrid
  - Clinica Universitaria de Navarra, Navarra
- University Hospital Zurich, Zurich, Switzerland
- United Kingdom (5):
  - Guy's Hospital, London
  - The Royal Marsden Hospital, London
  - Christie Hospital, Manchester
  - Nottingham University Hospitals NHS Trust, City Campus, Nottingham
  - Weston Park Hospital, Sheffield

REFERENCES:
- [Background] Bedikian AY, Agarwala SS, Gilles E, Itri L, Kay R, Garbe C. The AGENDA Study: A randomized, double-blind study of Genasense plus dacarbazine (DTIC) in chemotherapy-naïve subjects with advanced melanoma and low LDH. Pigment Cell Res. 2007;20:538 [Abstract T-26].
- [Background] Bedikian AY, Millward M, Pehamberger H, Conry R, Gore M, Trefzer U, Pavlick AC, DeConti R, Hersh EM, Hersey P, Kirkwood JM, Haluska FG; Oblimersen Melanoma Study Group. Bcl-2 antisense (oblimersen sodium) plus dacarbazine in patients with advanced melanoma: the Oblimersen Melanoma Study Group. J Clin Oncol. 2006 Oct 10;24(29):4738-45. doi: 10.1200/JCO.2006.06.0483. Epub 2006 Sep 11. PMID 16966688